CLINICAL TRIAL: NCT01652612
Title: Effects of Positive End-expiratory Pressure and Alveolar Recruitment on the Oxygenation and Respiratory Mechanics During One-lung Ventilation in the Supine Position
Brief Title: Positive End-expiratory Pressure and Alveolar Recruitment for One Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Yongseon Choi, assistant professor, Yonsei University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2011-0301
Record Dates: First submitted 2011-12-20; First posted 2012-07-30 (Estimated); Last update posted 2013-07-04 (Estimated); Status verified 2013-07

CONDITIONS: One Lung Ventilation
Keywords: positive end expiratory pressure

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): zero PEEP
- OLV strategy: PEEP (Experimental): 1. apply 8 cm H2O positive end expiratory pressure during one lung ventilation and until the end of surgery
  Interventions: Other: PEEP
- OLV strategy: PEEP followed by AR (Experimental): 1. alveolar recruitment strategy before one lung ventilation
  2. 8 cmH2O positive end expiratory pressure during one lung ventilation and until the end of surgery
  Interventions: Other: PEEP

INTERVENTIONS:
Other: PEEP — 8 cmH2O PEEP throughout the period of OLV and 2nd TLV
  Arms: OLV strategy: PEEP; OLV strategy: PEEP followed by AR

SUMMARY:
Hypoxia frequently develops during one lung ventilation in the supine position.The objective of this article is to study the impact of preemptive alveolar recruitment and subsequent positive end expiratory pressure on arterial oxygenation and lung mechanics during one lung ventilation in the supine position in patients undergoing thoracic surgery .

DETAILED DESCRIPTION:
outcome measures: respiratory parameters (Paw, Ppla, Compliance, Vd/Vt)and oxygenation parameters (PaO2, shunt fraction, Pa-AO2)

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* age: 20-75 years

Exclusion Criteria:

* moderate to severe impaired respiratory function,
* heart failure,
* patients' refusal

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
PaO2, number of patients with hypoxia (PaO2< 90mmHg) | participants will be followed for the duration of anesthesia, an expected average of 3 hours
  blood samplings after induction of anesthesia, 15 and 30 min after OLV, after the 2nd TLV

SECONDARY OUTCOMES:
intrapulmonary shunt | participants will be followed for the duration of anesthesia, an expected average of 3 hours
  blood sampling after induction of anesthesia, 15 and 30 min after OLV, after the 2nd TLV

CONTACTS AND LOCATIONS:
Overall Officials: Yongseon Choi, Principal Investigator — Assistant professor
Locations (1):
- Yong Seon Choi, Seoul, Seoul, South Korea